CLINICAL TRIAL: NCT05968079
Title: Performance Comparison Between Masimo W1™ and Apple Watch Series 8
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MACL0003
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Masimo W1™ and Apple Watch Series 8 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo W1™ and Apple Watch Series 8.
  Interventions: Device: Masimo W1™ and Apple Watch Series 8

INTERVENTIONS:
Device: Masimo W1™ and Apple Watch Series 8 — Noninvasive wearable health monitoring device

SUMMARY:
This study is also designed to compare the performance of Masimo W1™ and Apple Watch Series 8 against FDA cleared hospital grade pulse oximetry technology under desaturation conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 55 years of age.
* Subject is American Society Anesthesiologist status 1 (ASA I)
* Subject has a BMI between 18 and 35.
* Subject is able to read and communicate in English and understands the study and the risks involved.

Exclusion Criteria:

* Subject is currently taking any medications which in the opinion of the principal investigator would not be suitable for participation in the study.
* Subject is wearing nail polish that cannot be removed, gel nails, and/or acrylic nails that can interfere with study device's placement.
* Participants with conditions or skin abnormalities at or around site of sensor placement that could affect the placement on the sensor or prevent monitoring of physiological parameters during the study, such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown.
* Subject has participated in an investigational drug study within one month prior to the start of the study.
* Subject has failed the Allen's Test to confirm patency of the collateral artery.
* Subject is female with a positive pregnancy test, or is female and is unwilling to use effective birth control between the time of screening and study termination.
* Subject has a positive urine cotinine or drug test.
* Subject has a reported allergy to Lidocaine.
* Subject has clinically significant anemia or other hemoglobinopathy.
* Subject has a room air saturation of less than 95% by pulse oximetry.
* Subject has a clinically significant abnormal EKG.
* Subject has a clinically significant abnormal pulmonary function test via spirometry.
* Subject is intolerant to a breathing mask apparatus.
* Subject has a COHb greater than 3%, or MetHb greater than 2% verified by laboratory co-oximeter.
* Subject has another condition, which in the opinion of the principal investigator would not be suitable for participation in the study.
* Subject is unwilling or unable to provide informed consent or comply with the study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology and Physiology Laboratory (HPPL) - Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Masimo W1™ and Apple Watch Series 8
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 20 subjects were enrolled for the study
Arm/Group | Masimo W1™ and Apple Watch Series 8
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4
  Asian or Pacific Islander | 7
  Hispanic | 3
  White | 6

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Masimo W1™ and Apple Watch Series 8 in Determining SpO2 (Oxygen Saturation) Values in Subjects During Desaturation
Description: Accuracy will be determined by comparing Masimo W1™ SpO2 measurements and Apple Watch Series 8 SpO2 measurements with FDA-cleared pulse oximetry device SpO2 measurements and calculating the Arithmetic root mean square (ARMS) value. All values presented below for SpO2 (Bias, Precision and ARMS) are in units of %.
  The pairwise samples consist of paired SpO2 timing measurements from both the reference sensor, Masimo W1, and the Apple Watch.
Time Frame: 1-6 hours
Measure: Number; unit: Percent of oxygen saturated hemoglobin
Units Other Than Participants: Number of Pairwise Samples
Groups:
- Masimo W1™: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo W1™ and Apple Watch Series 8.
  Masimo W1™: Noninvasive wearable health monitoring device
- Apple Watch Series 8: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo W1™ and Apple Watch Series 8.
  Apple Watch Series 8: Noninvasive wearable health monitoring device
Arm/Group | Masimo W1™ | Apple Watch Series 8
Number analyzed (Participants) | 20 | 20
Number analyzed (Number of Pairwise Samples) | 398 | 398
Percent of oxygen saturated hemoglobin
  Clinical Bias | 0.4 | 0.8
  Precision | 1.9 | 2.0
  Arithmetic Root Mean Square (ARMS) | 2.0 | 2.2

2. Primary Outcome: Successful Read Rate for Motion Conditions Under Slow Desaturation for Masimo W1™ and Apple Watch Series 8
Description: This analysis examines the successful read rates for motion conditions during slow desaturation events for the Masimo W1™ and Apple Watch Series 8. The motion condition consists of a combined value representing three types of simulated motion: drinking, scratching the nose, and checking the time.
  Successful Read Rate = 1 - No Read Rate (Nf / Nspotcheck) x 100 (%) Nf = Number of Reads without Valid SpO2 Nspotcheck = Number of All Spot Checks
Time Frame: 1-6 hours
Measure: Number; unit: % of Successful Read Values
Units Other Than Participants: Number of Paired Spot Checks
Arm/Group | Masimo W1™ | Apple Watch Series 8
Number analyzed (Participants) | 20 | 20
Number analyzed (Number of Paired Spot Checks) | 400 | 400
% of Successful Read Values | 100 | 4.7

3. Primary Outcome: Detection Rate of Fast Desaturation Events Under Various Conditions for Masimo W1™ and Apple Watch Series 8
Description: Comparison of the detection rate of fast desaturation events under different conditions for the Masimo W1™ and Apple Watch Series 8. The first condition involves no motion, with the palm facing down and the Apple Watch in sleep mode, while the second condition involves no motion, with the palm facing sideways and manual spot checks performed on the Apple Watch. The goal is to evaluate the performance of both devices in detecting desaturation events under these varying circumstances.
  Detection Rate = (Nt / Ndesat) x 100 (%) Nt = Number of Detected Event by Test Device
  All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo W1™ and Apple Watch Series 8.
  Ndesat = Number of All Valid Fast Desaturation Events by Reference SpO2
Time Frame: 1-6 hours
Measure: Number; unit: Event Detection Rate (%)
Units Other Than Participants: Number of Valid Events
Arm/Group | Masimo W1™ | Apple Watch Series 8
Number analyzed (Participants) | 20 | 20
Number analyzed (Number of Valid Events) | 187 | 187
Event Detection Rate (%)
  Condition 1: No motion, palm facing down, Apple Watch in Sleep Mode | 100 | 7.4
  Condition 2: No motion, palm facing sideways, manual spot checks for Apple Watch | 100 | 24.7

ADVERSE EVENTS:
Time Frame: Through study completion, each subject's participation in the study was between 1-6 hours
Arm/Group | Masimo W1™ and Apple Watch Series 8
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT05968079/Prot_SAP_000.pdf